CLINICAL TRIAL: NCT05995028
Title: Safety and Efficacy of Universal 4SCAR7U T Cell Therapy Targeting CD7-positive Hematological Malignancies
Brief Title: Universal 4SCAR7U Targeting CD7-positive Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-23002
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Acute Lymphoblastic Lymphoma; Acute Myeloid Leukemia; NK Cell Lymphoma
Keywords: T-ALL; TCL; AML; NK lymphoma; Universal CAR T; CD7
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Universal 4SCAR7U cells to treat CD7-positive hematological malignancies (Experimental)
  Interventions: Biological: Universal CD7-specific CAR gene-engineered T cells

INTERVENTIONS:
Biological: Universal CD7-specific CAR gene-engineered T cells — Infusion of 4SCAR7U T cells

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of universal CAR T cells based on 4SCAR7U design against CD7-positive hematological malignancies using CD7 specific universal CAR T cells. The study also aims to learn more about the function of CD7 targeting CAR T cells and their persistence in patients of hematological malignancies.

DETAILED DESCRIPTION:
Hematological malignancies including B-, T-cell acute lymphoblastic leukemia (B-ALL, T-ALL), B and T cell lymphoma (BCL, TCL), natural killer cell lymphoma (NKL) and acute myeloid leukemia (AML) are aggressive diseases which may express the early T cell development molecule CD7.T-ALL represents 15% of childhood and 25% of adult ALL, and T-ALL patients are prone to early disease relapse and suffer from poor treatment outcomes. According to European Group for the Immunological Characterization of Leukemias (EGIL), the presence of cytoplasmic or membrane expression of CD3 defines T-ALL. Several immunophenotypic classifications have been proposed: (TI) the immature subgroup or pro-T-ALL is defined by the expression of CD7 and cCD3; (TII) pre-T-ALL also expresses CD2 and/or CD5 and/or CD8; (TIII) or cortical T-ALL shows CD1a positivity; and (TIV), mature T-ALL is characterized by the presence of surface CD3 and CD1a negativity.Over the past few years, T cells modified with lentiviral chimeric antigen receptor (CAR) gene have been studied in different clinical settings. CD7 is a T cell surface molecule that plays important role in T cell and B cell interaction in early lymphoid development, displays membrane expression early during T cell development before TCR rearrangement, and persists through terminal stages of T cell development, and has been a well-known marker for T-ALL. CD7 is considered a promising target for the treatment of T-ALL, TCL, AML and NKL. In this study, the study proposes to investigate an universal CD7 targeting CAR-T design, 4SCAR7U in combination with alternative targeting CAR-T cells as a new strategy to treat CD7-positive hematological malignancies.

The 4SCAR7U T cells are genetically engineered and manufactured in bulk amount that can be supplied off-the-shelf without being custom made from individual patients. The immediate availability of the CAR-T cells makes clinical treatment convenient and timely for rapid progressing disease or for highly immune suppressed patients. This application can be time- and cost-effective. This novel approach may also overcome problems of functionally defective autologous T cells. The purpose of this clinical trial is to assess the feasibility, safety and efficacy of the 4SCAR7U T cell product in hematological malignancies. Another goal of the study is to learn more about the function of this novel product and its persistence in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Confirmed expression of CD7 and additional surface antigens in the cancer cells by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV or hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
6. Previous treatment with any gene therapy products.
7. Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | 6 months
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Clinical response | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No